CLINICAL TRIAL: NCT04152525
Title: The Effect of Mindfulness-Based Education Given to Individuals With Substance-Use Disorder According to SelfEfficacy Theory on Self-Efficacy Perception
Brief Title: The Effect of Awareness-Based Education Given to Individuals With Substance Use Disorder on Self-Efficacy Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KaratayUB
Record Dates: First submitted 2019-09-30; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Nurse's Role; Self Efficacy; Substance Use Disorders
Keywords: Mindfulness; Theory
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single Blinded
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The mindfulness-based education programme that was conducted by the researcher and aimed at increasing self-efficacy in substance addicts was conducted within eight sessions, 2 days a week for 4 weeks.
  Interventions: Other: Psychoeducation
- control group (No Intervention): Routine care

INTERVENTIONS:
Other: Psychoeducation — The mindfulness-based education programme that was conducted by the researcher and aimed at increasing self-efficacy in substance addicts was conducted within eight sessions, 2 days a week for 4 weeks.
  Arms: experimental group

SUMMARY:
This study was conducted to determine the effect of mindfulness-based education given to individuals with substance-use disorder according to Self-Efficacy Theory on self-efficacy perception. Sample was 112 (ewperimental group: 56; control group: 56) alpha=0,05 and power=0,80 et the and of study. The experimental group recevied, prepared in accordance with mindfulness, self-efficacy theory psychoeducation program, the control group received routine care. Data were collected 2 times: pretest, 2 month after intervention (for experimental group) and 2 month after pretest (for control group).

DETAILED DESCRIPTION:
Substance use disorders are among the most important problems of our time. It has become a public health problem which is very common in developed and developing countries and affects the individual and the family as well as the society. Treatment of this problem, which leads to important disorders in many parts of individuals' lives, is quite difficult. Primary treatment is carried out by pharmacological methods. In cases where pharmacological methods are not sufficient, treatment is supported with psycho-social methods.

The aim is to identify the effect of mindfulness-based education, which is in accordance with self-efficacy theory, given to individuals who have substance abuse disorders.

The research was planned as a test model with pretest-posttest control groups. Individuals who have been diagnosed with substance abuse in the substance abuse clinic of Turgut Özal Medical Center, and at the Substance Abuse Treatment and Education Centre of Gaziantep 25 Aralık State Hospital formed the core of this study. The research was conducted between January 2018-May 2019. 112 patients, 56 in the treatment and 56 in the control group, participated in the study. Scientific research started after ethical approval. Mindfulness therapy was applied to experimental group patients. For the data collection, the Socio-Demographic Characteristics Questionnaire and Self-Efficacy scale were used. Kolmogorov-smirnov distribution test was used for normal distribution and Cronbach's alpha was used for internal consistency. Percentage, mean and standard deviation in evaluation of patients' demographic data, chi-square test in parametric cases in comparison of control variables of experimental and control groups, Fisher's exact test in non-parametric cases, t-test in dependent groups in comparison of mean scores of experimental and control groups, score in test and control groups in itself. t test was used in independent groups.

ELIGIBILITY:
Inclusion Criteria:

* To be able to communicate,
* 18 years and older,
* Diagnosis of substance use disorder according to the diagnostic criteria in DSM-V,
* No prior training in awareness therapy or self-efficacy theory,

Exclusion Criteria:

* Patients who actively use alcohol or psychoactive substances,
* Those who show withdrawal symptoms due to substance use disorder,
* Psychotic patients due to substance use
* Want to leave the work
* who cannot continue psychoeducation regularly
* low mental capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
self-efficacy score pretest for experimental group | first day of study
  self-efficacy level determined by pretest for the experimental group.The lowest score that can be obtained from the scale was evaluated as 23 and the highest as 115.The higher the score, the higher the level of self-efficacy.
self-efficacy score pretest for control group | first day of study
  self-efficacy level determined by pretest for the control group.The lowest score that can be obtained from the scale was evaluated as 23 and the highest as 115. The higher the score, the higher the level of self-efficacy.

SECONDARY OUTCOMES:
self-efficacy score posttest for experimental group | 2 month later
  Self-efficacy level increased in experimental group. The lowest score that can be obtained from the scale was evaluated as 23 and the highest as 115. The higher the score, the higher the level of self-efficacy.
self-efficacy score posttest for control group | 2 month later
  Self-efficacy level did not change in the control group. The lowest score that can be obtained from the scale was evaluated as 23 and the highest as 115. The higher the score, the higher the level of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: BERNA BAYIR, 1, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

REFERENCES:
- [Derived] Bayir B, Aylaz R. The effect of mindfulness-based education given to individuals with substance-use disorder according to self-efficacy theory on self-efficacy perception. Appl Nurs Res. 2021 Feb;57:151354. doi: 10.1016/j.apnr.2020.151354. Epub 2020 Aug 27. PMID 32907766